CLINICAL TRIAL: NCT06050551
Title: Comparison of Postoperative Small-bore Pigtail or Large-bore Chest Tube Placement After Uniportal Video-assisted Thoracoscopic Surgery for Postoperative Analgesia and Enhanced Recovery: a Randomized Controlled Trial.
Brief Title: Pigtail or Chest Tube Placement After Uniportal Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Yuan's General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Shuoying, medical doctor, attending physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221108B
Record Dates: First submitted 2023-08-26; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain, Acute; Post-Op Complication; Opioid Use, Unspecified; ERAS; Uniportal Video-Assisted Thoracic Surgery (VATS)
Keywords: post-operative analgesia; ERAS (Enhanced Recovery After Surgery); pigtail; chest tube
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14-Fr pigtail catheter after uniportal VATS (Experimental): smaller catheter used after uniportal VATS
  Interventions: Procedure: uniportal VATS
- 20-Fr chest tube after uniportal VATS (Other): routine management after uniportal VATS
  Interventions: Procedure: uniportal VATS

INTERVENTIONS:
Procedure: uniportal VATS — 1. elective uniportal VATS lung resection, pleural tumor removal or mediastinal lymph node biopsy, etc.
     (exclude the bil. operation, extended wound length over 5 cm, conversion to thoracotomy or multiportal VATS procedure, surgeon's decision for exclusion during operation.)
  2. thoracoscopic internal costal nerve block with 10 mL of 1% Ropivacaine at the end of the operation,
  3. routinely prescribed with oral Tramadol 37.5mg and Acetaminophen 325mg four times a day postoperatively and intravenous morphine as extra dose if need.

SUMMARY:
This study aims to figure out how small-bore pigtail catheter or large-bore chest tube for postoperative drainage impact on analgesic efficacy and actually enhance recovery postoperatively.

DETAILED DESCRIPTION:
Design A randomized controlled trial.

Setting The uniportal VATS has a small linear wound about 3 to 5 cm at only one intercostal space, mostly 4th or 5th. After elective thoracic surgery, the investigators routinely placed either one 14-Fr pigtail catheter or one 20-Fr chest tube for postoperative drainage.

The patients regularly receive thoracoscopic internal costal nerve block with 10 mL of 1% Ropivacaine at the end of the operation, and are routinely prescribed with oral Tramadol 37.5mg and Acetaminophen 325mg four times a day postoperatively and intravenous morphine as extra dose if need. The investigators check chest X ray on postoperative day one and try to remove the drainage tube soon if well lung expansion and ambulation without adverse events. Then the investigators will discharge this patient six hours later or the next day after drain removal smoothly.

Sample size determination and statistical analysis The patient number in one group will be calculated on the basis of significant pain relief and set as 33 patients with the following statistic parameter: α: 0.05 (type I error probability), power 0.8 (probability of correctly rejecting the null hypothesis), δ: 0.5 (difference in population means), σ: 1 (standard deviation of difference). The investigators added 20 % noncompliance rate and forty patients in each group (total eighty patients) will be included in this study.

Participants The investigators enrolled eighty consecutive adult patients, over 20 years old, undergoing elective uniportal VATS lung resection, pleural tumor removal or mediastinal lymph node biopsy, etc. The exclusion criteria are patient refusal, body mass index > 27 kg/m2, American society of anesthesiologists (ASA) grade above 3, contraindication to nerve block, allergy to analgesic agents, regular opioid used for chronic pain prior to this time surgery, anticipating postoperative patient control analgesia (PCA) before operation, surgeon's decision for exclusion during operation, conversion to thoracotomy or multiportal VATS procedure, postoperative intubation, postoperative intensive care unit admission.

Interventions Eighty adult patients, over 20 years old, were allocated randomly in a 1:1 ratio by computer-generated randomization to receive either one 14-Fr pigtail catheter or one 20-Fr chest tube for postoperative pleural drainage.

Measurement / Result The patient demographics, comorbidities, and thoracic surgical procedure, intra-operative blood loss, operative time, pathological results are reviewed.

The evaluation and measurement of primary and secondary outcomes are recorded by nurses or assistants at post-anesthetic care unit and ward. The independent samples t test, Chi-square test, Logistic Regression will be used for data analysis.

Primary outcome The resting and dynamic VAS (Visual Analogue Scale) while coughing and ambulation after operation 0, 2, 4, 8, 24, 48 hours are collected, as well as the postoperative nausea or vomiting episodes related to anesthesia or analgesia.

The investigators also record the first-time usage of intravenous morphine, cumulative intravenous morphine consumption in the first two postoperative days, and, if need, the additional analgesic agent or rescue analgesia requirement, such as patient controlled analgesia.

Secondary outcome The investigators record the function and daily amount of the pleural drainage, the interpretation of postoperative day one chest X ray, any attempts of additional pleural drain insertion or conversion to tube thoracotomy from pigtail catheter if need. In addition, the timing of chest tube removal, length of hospital stays, and surgical pulmonary complications or morbidity are also noted.

Conclusion The investigators will discover if the small-bore pigtail catheter placement would be equally or superiorly effective over analgesia and the following early recovery postoperatively after uniportal VATS, comparing to traditional chest tube. Then the protocol of minimally invasive thoracic operation will be revised and advanced.

ELIGIBILITY:
Inclusion Criteria:

- eighty consecutive adult patients undergoing elective uniportal VATS lobectomy

Exclusion Criteria:

- patient refusal, body mass index > 27 kg/m2, American society of anesthesiologists (ASA) grade above 3, contraindication to nerve block, allergy to analgesic agents, regular opioid used for chronic pain prior to this time surgery, anticipating postoperative patient control analgesia (PCA) before operation, surgeon's decision for exclusion during operation, conversion to thoracotomy or multiportal VATS procedure, postoperative intubation, postoperative intensive care unit admission.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The VAS (Visual Analogue Scale) | after operation 0, 2, 4, 8, 24, 48 hours
  resting and dynamic VAS (Visual Analogue Scale) while coughing and ambulation, the scale from "0" to "10", depending on the severity of pain. "0" means not painful, and "10" means the most pain in whole life.
morphine usage | in the first 24 hours after operation,
  cumulative intravenous morphine consumption
if there is any episodes of nausea or vomiting episodes that needs mediaction | after operation 0, 2, 4, 8, 24, 48 hours
  related to anesthesia or analgesia.

SECONDARY OUTCOMES:
pleural drainage from chest tube or pigtail, which was recorded by nurse. | after operation 24, 48, 72, 96 hours
  after uniportal VATS (Video-Assisted Thoracic Surgery)
if there is any timepoint for need of conversion to tube thoracotomy from pigtail catheter | after operation 24, 48, 72, 96 hours
  related to post-operative complications, such as massive pleural effusion, pneumothorax, unstable vital signs or respiratory failure
post-operative care after uniportal VATS (Video-Assisted Thoracic Surgery) | after operation 24, 48, 72, 96 hours
  the timing of chest tube removal and length of hospital stays

CONTACTS AND LOCATIONS:
Locations (1):
- Yuan's General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No